CLINICAL TRIAL: NCT06347328
Title: The Benefits of Posterior Joint Infiltration in Chronic Low Back Pain: a Randomised Study of the Benefits of Ultrasound-guided Infiltration Versus Unguided Infiltration. Prospective Randomised Study
Brief Title: The Benefits of Posterior Joint Infiltration in Chronic Low Back Pain
Acronym: InCHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-AOI-01
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low-back Pain
Keywords: infiltration; low back pain; facet joint; betametasone; pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-echo-guided infiltration (Active Comparator)
  Interventions: Procedure: non-echo-guided infiltration
- echo-guided infiltration (Experimental)
  Interventions: Procedure: echo-guided infiltration

INTERVENTIONS:
Procedure: echo-guided infiltration — the subjects will receive their injection in the ultrasound room. a glucocorticoid injection is given at the time of consultation, using anatomical ultrasound scan to guide needle placement
  Arms: echo-guided infiltration
Procedure: non-echo-guided infiltration — the subjects will receive their injection in the ultrasound room.
  a glucocorticoid injection is given at the time of consultation, using anatomical landmarks to guide needle placement.
  The investigator simulate an ultrasound scan with a film shown on the screen.
  Arms: non-echo-guided infiltration

SUMMARY:
Lumbar facet joints have been implicated in chronic low back pain in over 45% of patients with isolated chronic common low back pain.

Low back pain is the most common form of spinal pain, more chronic and severe than cancer pain. The annual prevalence of chronic low back pain ranges from 15% to 45% (one-off prevalence, 30%; lifetime prevalence, 54-80%). Because of this extremely high incidence, doctors from a wide range of specialities perform interventional techniques in a variety of settings.

Facet joints have long been recognised as a source of back pain. In 1911, Goldthwait first recognised their role as a potential source of back pain. In 1933, Ghormley introduced the term "facet syndrome", defining lumbosacral pain with or without radicular pain. Badgley later suggested that facet joints could be a primary source of pain independently of spinal nerve compression. They demonstrated the role of posterior facet joints (PFJs) in a large number of patients with low back pain whose symptoms were not caused by a herniated disc. The underlying physiological concept of the PJF was introduced by Hirsch et al in 1963. They demonstrated that injecting a hypertonic saline solution into the region of the facet joints caused pain.

The management of chronic low back pain due to zygapophyseal involvement (lumbar facet joints) consists primarily of conservative treatment. This is based on analgesics, anti-inflammatory drugs, physiotherapy and weight loss, where appropriate. Other non-surgical options may be proposed, including glucocorticoid injections into the facet joints. Glucocorticoid injections, which act by reducing inflammation, are commonly used in routine care to treat spinal pain. This pain may be due to a variety of pathologies, including discogenic or facet-related, or mixed, ligamentous or muscular, linked to a regional or global disorder of spinal statics. They are commonly used as a standard treatment for chronic spinal pain.

Traditionally, in routine clinical practice, if there is significant paravertebral contracture and the clinical signs point to posterior joint involvement, a glucocorticoid injection is given in the doctor's surgery at the time of consultation, using anatomical landmarks to guide needle placement. However, few studies have demonstrated the efficacy of anatomical marking for infiltration of posterior joints, notably Cohen et al. Sui's systematic review of the use of this technique.

With the advent of new imaging modalities such as ultrasound, more and more practitioners are turning to image-guided injections. To date, only the fluoroscopy-guided technique is considered reliable for facet joint infiltration.

In order to improve the clinical efficacy of the various interventional therapeutic solutions, some authors have supported the use of ultrasound guidance. Several studies have been published comparing ultrasound-guided infiltration and infiltration using anatomical location in the shoulder region, the iliopsoas and in epicondilitis. While ultrasound guidance in areas such as the iliopsoas or the shoulder seems useful, it has not yet been proven that guidance is advantageous in spinal areas, such as the facet joints.

To our knowledge, no randomised, methodologically sound study has yet been carried out to compare the benefit of ultrasound-guided infiltration versus infiltration with anatomical location.

The aim of our study is to show that ultrasound-guided zygoapophyseal infiltration is superior to anatomically-guided infiltration in terms of pain assessment.

DETAILED DESCRIPTION:
This is a multicentre, prospective, interventional study involving two groups of patients, randomised, blinded, category 2, at the Nice University Hospital, the Antibes University Hospital and the Cannes University Hospital. The control group will consist of patients receiving unguided infiltration. The experimental group will consist of patients receiving ultrasound-guided infiltration.

Inclusion and follow-up visits will be carried out at the following centres: Nice University Hospital, Antibes University Hospital and Cannes University Hospital. The infiltration (ultrasound-guided and non-ultrasound-guided) will be carried out by the rheumatologist sonographer at the Nice University Hospital only. The ultrasound will be performed by a trained rheumatologist using a low-frequency convex probe (1-8 MHz) and/or a linear probe (12-15 MhZ). The investigators will perform B-mode tracking in two perpendicular planes to locate the target. The probe will be positioned vertically about 3 to 4 cm to the left or right of the line of the spinous processes. The sonographic appearance of the spinous processes is easy to identify, as they form several 'bumps'. The injection will be carried out under strict aseptic conditions, with the lumbar puncture needle (20G) introduced in line with the probe at an angle of approximately 45° longitudinally to the axis of the posterior articular joints. The needle will be advanced under local anaesthetic using approximately 5 cc of 5% Xylocaine until contact with the bone, positioning and adapting the needle dynamically throughout the procedure. The symptomatic joint will be injected with 1 ml of betamethasone. The duration of the procedure (from disinfection to removal of the needle) will be recorded, as will the immediate post-gestational complications and finally the VAS of the pain felt by the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years
2. Isolated intermittent or continuous chronic low back pain resulting in functional disability;
3. Having undergone a CT scan or MRI of the lumbar spine, with the joint spaces of the lumbar facet visible, showing condensation or hypersignal of the posterior joints.
4. Somatic or non-radicular low back pain lasting at least three months;
5. Failure of conservative treatments, including physical therapy with exercises, chiropractic and pharmacological therapy;
6. Initial or recurrent lumbago lasting more than 3 months.
7. VAS pain greater than or equal to 4 on a scale of 0 to 10.

Exclusion Criteria:

1. Withdrawal of consent
2. Instability of the spine
3. Spondylodiscitis
4. Fracture of any location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change of pain progression | at inclusion, and three months after procedure
  The difference in pain progression between baseline and 3 months will be assessed using a visual analogue scale (0-100). The VAS is graduated from 0 to 100 mm, with 0 = no pain and 100 = maximum pain perceived in the 48 hours preceding the consultation, as recommended by the OARSI in osteoarthritis on pain assessment. The pain VAS will be assessed at rest, at night and during activities. This will be documented at the start of the study, and three months later, using the VAS and the remission rate (VAS < 4).

SECONDARY OUTCOMES:
measure function state by EIFEL questionnaire | at inclusion and 3 months after procedure
  In french "Echelle d'Incapacité Fonctionnelle pour l'Evaluation des Lombalgies" (EIFEL) questionnaire is a Functional Disability Scale for the Assessment of Low Back Pain.
  The questionnaire is composed of 24 sentences to describe the patient's physical condition. The maximal value is 24, means a very disabling functional disability. Higher scores mean a worse outcome.
  The difference in the evolution of the EIFEL questionnaire between baseline and 3 months compared between the two groups will be measured.
  The EIFEL index is a french translation of the Rolland Morris questionnaire and has been validated for acute low back pain. It explores disability by combining handicap, impairment and incapacity.
measure function state by ODI questionnaire | at inclusion and 3 months after procedure
  Evaluation of the difference in patients' functional status using the Oswestry Disability Index (ODI) between baseline and 3 months, compared between the two groups.
  The Oswestry Low Back Pain Disability Questionnaire is used to measure the extent of pain-induced functional limitations in people with low back pain. The questionnaire provides the user with details of the general day-to-day functioning of the low back pain patient. Six response options are available for the following items: pain intensity, personal care (washing, dressing), lifting objects, moving around, sitting or standing, sleeping, sex life, social life, and travel/transportation. The first response option (score 0) denotes the absence of pain-related restrictions, while the sixth response option (score 5) denotes the greatest perceived restriction of an activity caused by pain.
pain evaluation by VAS scale | at 30 minutes , one month and two months after the procedure
  The VAS is graduated from 0 to 100 mm, with 0 = no pain and 100 = maximum pain perceived.The pain VAS will be assessed at rest, at night and during activities. This will be documented at t 30 minutes after the procedure, one month, two months later, using the VAS and the remission rate (VAS < 4).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de NICE, Nice, CHU de Nice
  - Ch Cannes, Cannes